CLINICAL TRIAL: NCT01383434
Title: A Phase II Trial of Myeloablative Conditioning and Transplantation of HLA-matched, Partially HLA-mismatched, HLA-haploidentical or Matched Unrelated (MUD) Bone Marrow for Patients With Refractory Severe Aplastic Anemia
Brief Title: Bone Marrow Transplant Trial for Patients With Refractory Severe Aplastic Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: New revised SAA BMT study opened to take over this study
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J10117; NA_00042991 (Other: The Johns Hopkins University)
Record Dates: First submitted 2011-06-22; First posted 2011-06-28 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Bone Marrow Transplant — Matched sibling, haploidentical or matched unrelated donor bone marrow transplant following chemotherapy

SUMMARY:
Patients with severe, refractory aplastic anemia have a severe, life threatening disease in their bone marrow. Refractory disease means that disease has come back or not responded after receiving one or more immunosuppressive treatments. High dose chemotherapy followed by bone marrow transplantation (BMT) has been used to treat blood diseases like aplastic anemia but complications from Graft vs Host disease (GVHD) and graft failure have limited the survival for those patients.

Another study done here at Johns Hopkins has shown that in patients with other diseases (blood cancers) some immunosuppressive drugs given after the BMT has decreased how often patients had complications of GVHD and engraftment failure.

This research is being done to find if this approach will help patients with aplastic anemia who have failed other treatments will have better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have refractory or relapsed SAA following treatment with one or more immunosuppressive regimens.
* Age 6 months - 70 years
* Patients must meet medical criteria for myeloablative BMT
* Patients or their parents/guardians and donors must be able to sign consent forms.
* Patients must be geographically accessible and willing to participate in all stages of treatment.

Exclusion Criteria:

* Poor cardiac function: left ventricular ejection fraction <45% as determined by MUGA or ECHO.
* Poor pulmonary function: FEV1 and FVC <50% predicted.
* Poor renal function
* Positive leukocytotoxic crossmatch
* Women of childbearing potential who currently are pregnant (Β-HCG+) or who are not practicing adequate contraception
* Uncontrolled viral, bacterial, or fungal infections

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To estimate the overall survival (OS) at 1 year following HLA-matched, Partially HLA-mismatched, HLA-haploidentical or matched unrelated Bone Marrow for Patients with Refractory Severe Aplastic Anemia | 1 year
To estimate the event-free survival (EFS) at 1 year following HLA-matched, Partially HLA-mismatched, HLA-haploidentical or matched unrelated Bone Marrow for Patients with Refractory Severe Aplastic Anemia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Brodsky, MD, Principal Investigator — The Johns Hopkins University; Amy Dezern, MD, Principal Investigator — The JOhns Hopkins Sydney Kimmel Comprehensive Cancer Center
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States